CLINICAL TRIAL: NCT01862107
Title: Cerebrospinal Fluid Collection and Repository Storage
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to limited resources and declining participation.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130140; 13-N-0140
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2024-06

CONDITIONS: Nervous System Diseases
Keywords: Biomarkers; Immune Responses; Lumbar Puncture; Neurological Diseases; Novel Pathogens; Natural History
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Any healthy volunteer getting a lumbar puncture done for either clinical care or research purposes.
- Patient: Any patient getting a lumbar puncture done for either clinical care or research purposes.

SUMMARY:
Background:

- Cerebrospinal fluid (CSF) is the liquid around the brain and spinal cord. Many diseases can only be diagnosed by examining the CSF. A lumbar puncture is used to collect and test CSF. Once someone is already having a lumbar puncture, a small extra amount of CSF can be collected at the same time. This fluid can be used to study brain, nerve, and related health issues. Researchers want to collect CSF and blood samples from people who are scheduled to have a lumbar puncture.

Objectives:

- To collect cerebrospinal fluid and blood samples from individuals who are having a lumbar puncture.

Eligibility:

- Individuals between 2 and 100 years of age who are scheduled to have a lumbar puncture for clinical or research purposes.

Design:

* Participants will have a lumbar puncture for clinical or research purposes.
* During the procedure, an additional sample of CSF will be collected. They will also provide a blood sample, if one is not taken at the time of the procedure.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
In this study we are planning to establish a repository of cerebrospinal fluid (CSF), serum, and plasma. We are planning to collect a small amount of additional CSF and blood on subjects who are already going to have a lumbar puncture as part of their research or clinical care at the National Institutes of Health (NIH). This will allow us to study whether there is an association between neurological diseases and biomarkers, help identify novel pathogens infecting the central nervous system, and better enable us to understand the immune response to infections under future protocols. CSF and blood as well as clinical data associated with the samples will be stored securely.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:
* Subjects (patients and healthy volunteers) 2 years of age and older identified to undergo LP for research or for clinical care purposes at the NIH Clinical Center.

SUBJECT EXCLUSION CRITERIA:

-Subjects (patients and healthy volunteers) with the inability to provide informed consent either directly or via a legally authorized representative.

Inclusion of Vulnerable Subjects - Research Involving Adults Who Are Or May Be Unable To Consent:

-The risks to all subjects involved in this research project are no more than minimal risk as we are only collecting additional CSF and plasma during a LP procedure that is already being performed under a separate research protocol or as a clinically indicated procedure. At the time of the LP it will already be determined if the subject is able to give informed consent and if not a legally authorized representative will have been appointed who will decide if the additional CSF and plasma can be obtained from the individual.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study is a collection of additional CSF from any patient getting a lumbar puncture done for either clinical care or research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to create a repository of CSF and matched serum and plasma samples. | ongoing
  Repository of CSF and matched blood.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuntz KM, Kokmen E, Stevens JC, Miller P, Offord KP, Ho MM. Post-lumbar puncture headaches: experience in 501 consecutive procedures. Neurology. 1992 Oct;42(10):1884-7. doi: 10.1212/wnl.42.10.1884. PMID 1407567
- [Background] Silverberg GD, Heit G, Huhn S, Jaffe RA, Chang SD, Bronte-Stewart H, Rubenstein E, Possin K, Saul TA. The cerebrospinal fluid production rate is reduced in dementia of the Alzheimer's type. Neurology. 2001 Nov 27;57(10):1763-6. doi: 10.1212/wnl.57.10.1763. PMID 11723260
- [Background] Ebinger F, Kosel C, Pietz J, Rating D. Headache and backache after lumbar puncture in children and adolescents: a prospective study. Pediatrics. 2004 Jun;113(6):1588-92. doi: 10.1542/peds.113.6.1588. PMID 15173478
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-N-0140.html